CLINICAL TRIAL: NCT02721407
Title: A Phase I Study of Anti-CD22:TCRz:4-1BB T-cells in Patient With CD22-Positive Recurrent Lymphoma That is Resistant or Refractory to Prior Anti-CD22:TCRz:CD28 Immunotherapy
Brief Title: Anti-CD22 CAR-T Therapy for CD19-refractory or Resistant Lymphoma Patients
Acronym: MendCART
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Qingzhu Jia, M.D., Director of Department of Cancer, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CD22CART
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Stage III/IV Adult Diffuse Large Cell Lymphoma; Stage III/IV Follicular Lymphoma; Stage III/IV Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, Mantle-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Anti-CD22 CAR-T (Experimental): Administrated with CD22.CAR-T cells on day 0,1,2 in the lympho-depleted patients
  Interventions: Drug: Retroviral vector-transduced autologous T cells to express CD22-specific CARs

INTERVENTIONS:
Drug: Retroviral vector-transduced autologous T cells to express CD22-specific CARs

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-CD22:TCRz:4-1BB chimeric antigen receptor (CAR)-modified T (CAR-T) cells in treating recurrent patients with refractory or resistant lymphoma to anti-CD19:TCRz:CD28 CAR-T cells. Recently, cancer immunotherapy, treatments aiming to arm patients with immunity specifically against cancer cells, has emerged as a promising therapeutic strategy. Among the many emerging immunotherapeutic approaches, clinical trials utilizing CARs against B cell malignancies have demonstrated remarkable potential. CARs combine the variable region of an antibody with T-cell signaling moieties to confer T-cell activation with the targeting specificity of an antibody. Thus, CARs are not MHC-restricted so they are not vulnerable to MHC down regulation by tumors. However, defined by the recession of evaluable lesions, the persistence and efficacy of CAR-T cells are still restricted by the "target" selection. Previous clinical studies largely utilized CD19 for the in vivo targeting of CAR-T cells, which preferentially become refractory or resistant due to the heterogeneity of lymphoma. This clinical investigation is to test a hypothesis whether anti-CD22 CAR-T cells work more effective in lymphoma patients refractory or resistent to anti-CD19:TCRz:CD28 CAR-T cells.

DETAILED DESCRIPTION:
Primary Objectives

1. To determine the safety of CD22.CAR-T cells in lymphoma patients refractory or resistent to anti-CD19:TCRz:CD28 CAR-T cells
2. To determine in vivo dynamics and persistency of CD22.CAR-T cells.

Secondary Objectives

1. To determine the feasibility of CD22.CAR-T cells in lymphoma patients refractory or resistent to anti-CD19:TCRz:CD28 CAR-T cells
2. To determine in vivo dynamics and persistency of CD22.CAR-T cells.
3. To assess the intratumoral infiltration of CD22.CAR-T cells.
4. To correlate the subsets and differentiation of CD22.CAR-T cells to observed anti-tumor efficacy

ELIGIBILITY:
Inclusion Criteria:

1.18 Years to 70 Years, Male and female;

2.Expected survival > 12 weeks;

3.Performance score 0-2;

4.Histologically confirmed as CD19-positive lymphoma and who meet one of the following conditions;

* Patient receive at least 2-4 prior combination chemotherapy regimens (not including single agent monoclonal antibody therapy) and fail to achieve CR; or have disease recurrence; or not eligible for allogeneic stem cell transplantation; or disease responding or stable after most recent therapy but refused further treatment;
* Disease recurrence after stem cell transplantation;
* Diagnosis as lymphoma, but refuse conventional treatment such as chemotherapy, radiation, stem cell transplantation and monoclonal antibody therapy

  5.Creatinine < 2.5 mg/dl;

  6.ALT/AST < 3x normal;

  7.Bilirubin < 2.0 mg/dl;

  8.Adequate venous access for apheresis, and no other contraindications for leukapheresis;

  9.Take contraceptive measures before recruit to this trial;

  10.Written voluntary informed consent is given.

  11.Refractory ot resistant to prior anti-CD19 CAR-Ts

  12.At least one evaluable CD22-positive recurrent lesion, confirmed by two independent pathologist.

Exclusion Criteria:

1. Patients with symptoms of central nervous system
2. Accompanied by other malignant tumor
3. Active hepatitis B or C, HIV infection
4. Any other diseases could affect the outcome of this trial
5. Suffering severe cardiovascular or respiratory disease
6. Poorly controlled hypertension
7. A history of mental illness and poorly controlled
8. Taking immunosuppressive agents within 1 week due to organ transplantation or other disease which need long-lasting administration
9. Occurrence of unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events 30 days prior to assignment
10. Reaching a steady dose if receiving anticoagulant therapy before assignment
11. Female study participants of reproductive potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
12. Pregnant or lactating women
13. Subject suffering disease affects the understanding of informed consent or comply with study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 4.0 | 4 Weeks

SECONDARY OUTCOMES:
Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm | 8 Weeks
Duration of CAR-positive T cells in circulation | 6 months
Total number of CAR-positive T cells infiltrated into lymphoma tissue | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes